CLINICAL TRIAL: NCT04401735
Title: Effects and Safety of PDRN (Polydeoxyribonucleotide) for Patient With Lumbar Spinal Stenosis Compared With Normal Saline in Randomized Placebo-Controlled Comparative Pilot Study
Brief Title: Effects and Safety of Epidural PDRN vs. Placebo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Pyung-Bok Lee, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUBHPAIN
Record Dates: First submitted 2020-05-11; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Spinal Stenosis Lumbar
MeSH Terms: interventions — Polydeoxyribonucleotides; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Polydeoxyribonucleotide (Experimental): Polydeoxyribonucleotide(PDRN) 5.625mg/3ml
  Interventions: Drug: Polydeoxyribonucleotides
- Polydeoxyribonucleotide, Placebo (Experimental): Polydeoxyribonucleotide(PDRN) 5.625mg/3ml Placebo (Normal saline)
  Interventions: Drug: Polydeoxyribonucleotides; Drug: Normal saline
- Placebo (Placebo Comparator): Placebo (Normal saline)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Polydeoxyribonucleotides — PDRN injection to epidural space
  Arms: Polydeoxyribonucleotide; Polydeoxyribonucleotide, Placebo
Drug: Normal saline — Normal saline
  Arms: Placebo; Polydeoxyribonucleotide, Placebo

SUMMARY:
This is a single-center, randomized, double-blind clinical study to assess the clinical application and outcomes with epidural PDRN versus Normal saline injection in patients with spinal stenosis.

DETAILED DESCRIPTION:
Patients who are already planning to receive an Transforaminal epidural block from their clinician will be approached by study members on the day of their injection. If enrolled, the patients will be contacted every 2 weeks for 4 weeks to determine the severity of pain and degree of pain relief from the injection.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults aged between 19-80 years old
* 2. Radiological confirmation of spinal stenosis on MRI
* 3. Neurogenic claudication greater thanVAS 4 of due to spinal stenosis
* 4. Follow-up possible during 3 months the clinical trial

Exclusion Criteria:

* Not able to comply fully with the protocol, including treatment, follow-up or study procedures
* pregnant or feeding women
* Alcohol/drug abuse
* Anticoagulant medication

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale(VAS) | 12 weeks post - injection
  This is in pain measurement ranging from 0 when no pain to 10 when there is severe pain(low back pain)

SECONDARY OUTCOMES:
visual analogue scale(VAS) | 4, 8 weeks post - injection
  This is in pain measurement ranging from 0 when no pain to 10 when there is severe pain(low back pain)
CGI(Clinicians Global Impression) | 4, 8 weeks post - injection
  7 point scale that requires the clinician to assess how much the patient's illness has improved(grade 0) or worsened(grade 7) relative to a baseline state at the beginning of the intervention.
treadmill test | 8 weeks post - injection
  walking distance

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university Bundang hospital, Seongnam, Kyoung-ki-do, South Korea